CLINICAL TRIAL: NCT05438511
Title: A Formative Evaluation For Improving Breast Cancer Hormone Receptor Testing in Tanzania
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-480
Record Dates: First submitted 2022-06-17; First posted 2022-06-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: breast cancer hormone receptor testing; breast cancer testing; GeneXpert STRAT4; Memorial Sloan Kettering Cancer Center; 21-480
MeSH Terms: conditions — Breast Neoplasms | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants of focus groups: Breast cancer survivor, patient advocate or key healthcare personnel including hospital and laboratory leaders, pathologists, laboratory scientists and technicians, oncologists, nurses, and surgeons
  Interventions: Behavioral: Focus group; Behavioral: Organizational Readiness for Implementing Change

INTERVENTIONS:
Behavioral: Focus group — A semi-structured focus group discussion guide will be developed with question probes that cover 1) contextual factors, 2) barriers to implementation, and 3) facilitators to implementation, with secondary probing questions.
Behavioral: Organizational Readiness for Implementing Change — measures the extent to which organizational members are prepared to implement organizational change. The ORIC tool asks participants to rate their level of agreement with 12 statements pertaining to organizational readiness for change (change commitment and change efficacy) on a 5-point Likert Scale.
  Other Names: ORIC tool

SUMMARY:
The purpose of this study is to learn more about the challenges with breast cancer diagnosis in Tanzania and the support available to improve this process.

ELIGIBILITY:
Participant Inclusion Criteria for interviews and focus group discussions (Aims 1 and 2):

* Breast cancer survivor, patient advocate or key healthcare personnel

  * Key healthcare personnel are defined as hospital and laboratory leaders, pathologists, laboratory scientists and technicians, oncologists, nurses, and surgeons, with:
  * >12 months of employment at the affiliated institution
  * Administrative or clinical involvement in the delivery of breast cancer care services.
* Age 18 years and above
* Permanent residents or citizens of Tanzania
* Participant and/or LAR willing and able to consent
* Fluent in Swahili and/or English by self-report

Participant Exclusion Criteria:

* Key stakeholder not residing at their particular institutions during data collection will be excluded.

Eligibility criteria for Chart Reviews (Aim 1)

Inclusion Criteria for chart review:

* Age 18 years and above
* Permanent residents or citizens of Tanzania
* Received breast cancer diagnosis

Exclusion Criteria for chart review:

* Participants less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aim 1: We will use purposeful sampling to select the study participants of 70 participants. The representative participants from the following groups will be identified: hospital and laboratory leadership, pathologists, laboratory scientists and technicians, oncologists, surgeons, nurses, and patient survivors/patient advocates. With the exception of patient survivors and patient advocates, each focus group discussion will have only 1-2 representatives from a particular stakeholder group. Stakeholders will be adults, must have already completed their clinical or laboratory training, and have at least one year of clinical experience in breast cancer care. Patient survivors and patient advocates will be interviewed separately, and must be adults and with a prior diagnosis of breast cancer.
  Aim 2: Participants that were recruited in Aim 1 will be offered the opportunity to participate in follow up interviews to brainstorm implementation strategies.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Identify barriers for breast cancer diagnosis in Tanzania. | 1 year
  Depending on results of this initial evaluation, either additional data will be collected, or if successful, will use the data to begin identifying context-specific implementation strategies using the 'Implementation Mapping' framework1 . In a future protocol, these data will then be used to develop a strategy for an intervention that addresses urgent evidence-to-practice gaps in breast cancer diagnosis in Tanzania, and has the potential to help patients with breast cancer in sub-Saharan Africa (SSA) in the future. The collection of this key information will assist us and our collaborators to generate background data that can be used to develop and/or complement future clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Ng, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org